CLINICAL TRIAL: NCT03639220
Title: Photobiomodulation Therapy Combining Laser Diodes, Light-emitting Diodes in Exercise Capacity Assessed by 6MST in Patients With COPD - A Crossover, Randomized, Triple-blinded, Placebo-controlled Clinical Trial
Brief Title: Photobiomodulation Therapy in Exercise Capacity Assessed by 6MST in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: COPD_PBMT
Record Dates: First submitted 2018-08-08; First posted 2018-08-21 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Randomization will be held by drawing lots, which we use to determine whether the active combination of superpulsed lasers, LEDs, comprising the PBMT or the placebo will be given during the first session. During the second session, participants will receive the opposite treatment compared to their first session. Randomization labels will be created using a randomization table at a central office where a series of sealed, opaque, and numbered envelopes ensured confidentiality.
Who Masked: Participant, Investigator
Masking Description: A participating researcher who programmed the PBMT device (Multi Radiance Medical™, Solon, OH) based on the randomization results performed the randomization. He will be instructed not to inform the participants or other researchers of the PBMT dose (active or placebo). Thus, the researcher who performed the PBMT will be blinded to the dose administered to the participants. To further maintain blinding, participants used opaque goggles to prevent them from seeing whether a light will be irradiated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Photobiomodulation Therapy (PBMT) active (Active Comparator): Participants received active PBMT
  Interventions: Device: Photobiomodulation Therapy (PBMT)
- Photobiomodulation Therapy (PBMT) placebo (Placebo Comparator): Participants received placebo PBMT
  Interventions: Device: Photobiomodulation Therapy (PBMT)

INTERVENTIONS:
Device: Photobiomodulation Therapy (PBMT) — Phototherapy device - Multi Radiance Medical™ (Solon, OH, EUA)

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by dyspnea, as well as musculoskeletal and systemic manifestations. Photobiomodulation therapy (PBMT) with use of low-level laser therapy (LLLT) and/or light emitting diode therapy (LEDT) is an electrophysical intervention that has been found to minimize or delay muscle fatigue. The aim of this study is to evaluate the acute effect of PBMT with combined use of lasers diodes, light emitting diodes (LEDs), on muscle performance, exercise tolerance and metabolic variables during the 6-minute stepper test (6MST) in patients with COPD. Twenty-one patients with COPD will completed the 6MST protocol over 2 weeks, with 1 session per week. PBMT or placebo (PL) will be performed before each 6MST (17 sites on each lower limb, with a dose of 30 J per site, using a cluster of 12 diodes: 4 × 905 nm super-pulsed laser diodes, 4 × 875 nm infrared LEDs, and 4 × 640 nm red LEDs; Multi Radiance Medical™, Solon - OH, USA). Patients will be randomized into two groups before the test according to the treatment they will receive. Assessments will be performed before the start of each protocol. The primary outcomes are oxygen uptake and number of steps, and the secondary outcome are perceived exertion (dyspnea and fatigue in the lower limbs).

DETAILED DESCRIPTION:
All patients will have a diagnosis of COPD according to the global initiative for chronic obstructive lung disease (GOLD) criteria. The patients will be at a stable phase of the disease, indicated by a lack of change in medical therapy (including oral steroids) or an exacerbation of symptoms in the preceding 4 weeks. Patients with other known severe chronic diseases, including cardiac, neuromuscular, or orthopedic disorders, will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients
* Patients are at a stable phase of the disease

Exclusion Criteria:

* Patients with cardiac diseases
* Neuromuscular diseases
* Orthopedic disorders

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-09-02 (Actual)

PRIMARY OUTCOMES:
The primary outcomes are oxygen uptake | 1 week
  The 6MST aims to measure the oxygen uptake performed on a stepper in 6 minutes. During the 6MST, the rates of oxygen consumption (VO2) will be measured using a gas analyzer.

SECONDARY OUTCOMES:
The secondary outcomes are number of steps | 1 week
  The 6MST aims to measure the number of steps performed on a stepper in 6 minutes. A step was defined as a single complete movement of raising one foot and putting it down. The stepper will be placed on the ground facing a wall to allow patients to maintain their balance by placing their fingers on the wall. The step height is set at 20 cm. The number of steps performed in 6 minutes will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Miranda, PhD, Principal Investigator — Nove de Julho University
Locations (1):
- Laboratory of Phototherapy in Sports and Exercise, Universidade Nove de Julho (UNINOVE), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No